CLINICAL TRIAL: NCT04784234
Title: A Prospective Randomized Controlled Trial of GlaucoCetin vs Placebo in Glaucoma Patients With Visual Field Loss.
Brief Title: Vision Preservation and Restoration Following a 6 Month Trial of GlaucoCetin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: company was bought and discontinued producing supplement
Sponsor: Wills Eye (Other)
Collaborators: Guardian Health Sciences, Inc. (Unknown)
Responsible Party: Principal Investigator, Natasha Nayak Kolomeyer, MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB #2020-145
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Primary Open Angle Glaucoma
Keywords: primary open angle glaucoma; visual field loss; vision enhancement; GlaucoCetin; Neuroprotection
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Study aims to enroll 50 patients within each intervention arm (GlaucoCetin vs Placebo). Within the intervention arm there will be one group with Central visual field defects and one group with Peripheral visual field defects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking of GlaucoCetin and identical Placebo was provided by Guardian Health Sciences, Inc. Labeling has been conducted by non-clinical study team personnel in Glaucoma Research Center at Wills Eye Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GlaucoCetin Peripheral Group (Active Comparator): Primary Open Angle Glaucoma participants who meet inclusion exclusion criteria with peripheral visual field loss will be randomly assigned GlaucoCetin, a medical food in capsule form.
  Interventions: Dietary Supplement: GlaucoCetin
- Placebo Peripheral Group (Placebo Comparator): Primary Open Angle Glaucoma participants who meet inclusion exclusion criteria with peripheral visual field loss will be randomly assigned a placebo, with no nutritional value, in capsule form.
  Interventions: Other: Placebo
- GlaucoCetin Central Group (Active Comparator): Primary Open Angle Glaucoma participants who meet inclusion exclusion criteria with central visual field loss will be randomly assigned GlaucoCetin, a medical food in capsule form.
  Interventions: Dietary Supplement: GlaucoCetin
- Placebo Central Group (Placebo Comparator): Primary Open Angle Glaucoma participants who meet inclusion exclusion criteria with central visual field loss will be randomly assigned a placebo, with no nutritional value, in capsule form.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: GlaucoCetin — GlaucoCetin, a medical food in capsule form, is FDA regulated and includes ingredients that have been shown to support and protect mitochondrial function of retinal ganglion cells. GlaucoCetin consists of a mixture of Curcumin, N-Acetyl Cysteine, Ginkgo Biloba Extract, Alpha-lipoic Acid, Citicoline, Grape Seed Extract, Green Tea Extract, and Coenzyme Q10. Additional ingredients include L-Taurine, Niacinamide, Biotin, Natural Astaxanthin, Fisetin, Quercetin, Luteolin, Proprietary Dragonberry Flavor Complex, Monk Fruit, Bitter Blocker Natural Flavor, Citric Acid, Silica Dioxide, Fibersol-2, L-Leucine. Many of these are known anti-inflammatory and antioxidant ingredients. A 6 month supply of capsules, made for this study, will be provided at randomization with the following instructions: Take 6 capsules by mouth once daily with food.
  Arms: GlaucoCetin Central Group; GlaucoCetin Peripheral Group
Other: Placebo — The placebo is an identical capsule to the GlaucoCetin, made for this study, with no nutritional value. A 6 month supply of capsules will be provided at randomization with the following instructions: Take 6 capsules by mouth once daily with food.
  Arms: Placebo Central Group; Placebo Peripheral Group

SUMMARY:
This study is looking at changes in vision and visual function before and after a six month trial of a daily medical food called GlaucoCetin, formulated with ingredients to support and protect the optic nerve cells. Open angle glaucoma patients will be randomized to receive either a placebo or the medical food for 6 months. We hope to learn if this medical food can improve the vision of our glaucoma patients and to report the findings obtained to the general public.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the improvement in vision and visual function during a 6 month trial of GlaucoCetin versus placebo in patients with open angle glaucoma. The secondary objective is to evaluate change in quality of life, electrophysiologic response, and contrast sensitivity.

Procedures involved during participation include review of medical/ocular history, best corrected visual acuity, multiple Humphrey visual field testing 24-2 and 10-2 , Octopus G-Top, pattern electroretinogram (PERG), ocular coherence tomography (OCT), ocular coherence tomography angiography (OCTA), intraocular pressure (IOP), contrast sensitivity testing (CSV-1000), corneal hysteresis, biomicroscopy, fundus exam, disc photos, and serum testing.

To evaluate quality of life, included in testing is Compressed Assessment of Ability Related to Vision (CAARV). Responses to multiple surveys regarding vision related quality of life (GQL-15, Glaucoma Symptom Scale (GSS), National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25)) and diet (NHANES Dietary Screener) will be captured. Number of daily steps will be monitored at 2 intervals during the study using pedometers.

ELIGIBILITY:
Inclusion Criteria:

* Age of 40 to 80 years
* Bilateral open angle glaucoma with reliable visual field defects (at least one eye with mean deviation (MD) between -4.00 to -10.00 decibels (dB) on Humphrey Visual Field 24-2.

  * Group 1 (Peripheral): meets 1 hodapp-parrish-anderson (HPA) criteria for defect (3 contiguous points depressed on the pattern standard deviation (PSD) p <5%, one of which is depressed at p <1% level), and does not meet below paracentral criteria for Group 2.
  * Group 2 (Central): at least 1 paracentral point repeatedly depressed at p<1% on 24-2. Also meets the HAP criteria outlined above.
* Visual acuity 20/40 or better in each eye
* Intraocular Pressure (IOP) controlled at 2 measurements >3 months
* Clear media

Exclusion Criteria:

* Known bleeding disorder
* History of epilepsy or on anti-seizure medication
* Uncontrolled hypertension or diabetes
* Uncontrolled IOP
* Eye pathology leading to inaccurate IOP measurement
* Visually significant retinal pathology affecting vision in past or active (such as diabetic retinopathy or age related macular degeneration)
* Non-glaucomatous optic neuropathy
* Visually significant cataract (worse then 2+ cataract, or what is determined visually clinically significant by physician)
* History of ocular trauma
* Selective laser trabeculoplasty or laser procedure within past 3 months
* Cataract surgery within past 3 months
* Incisional glaucoma surgery within 6 months
* Current use of nitroglycerin
* Current use of antiplatelet therapy besides aspirin (such as clopidogrel) or anticoagulation (such as warfarin)
* Current use of systemic steroids or immunomodulating agents such as methotrexate.
* Sensitivity or allergy to any ingredients in GlaucoCetin: Curcumin, L-Taurine, N-Acetyl Cysteine, Niacinamide, Ginkgo Biloba, Lipoic Acid, Citicoline, Grape Seed Extract, Green Tea Leaf Extract, Coenzyme Q10, Biotin, Natural Astaxanthin, flavonoid complex containing Fisetin, Quercetin, and Luteolin
* Recent change in systemic medications or vitamins
* Use of Biotin, Ginkgo Biloba, Citicoline within past 3 months (or any other Glaucocetin ingredients within 1 month)
* Unreliable visual fields
* Unwilling to take supplement or placebo for 6 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Visual Field Mean Deviation | 3 hour examinations during a 6 month period
  Improvement in visual field mean deviation, measured in decibels, will be compared before, during and after a 6 month trial of daily GlaucoCetin vs Placebo capsules.

SECONDARY OUTCOMES:
Perceived Quality of Life Improvement | 20 minute questionnaires during a 6 month period
  Improvement in participants perceived vision-related quality of life (GQL-15, Glaucoma Symptom Scale (GSS)
Perceived Quality of Life Improvement measured by National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25) | 20 minute questionnaires during a 6 month period
  Improvement in participants perceived vision-related quality of life ( National Eye Institute Visual Function Questionnaire 25 (NEI VFQ-25))

CONTACTS AND LOCATIONS:
Overall Officials: Natasha N Kolomeyer, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Glaucoma Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No